CLINICAL TRIAL: NCT03295539
Title: MulticentRe pOst-market exPeriencE With the INdigo Thrombectomy System for the Treatment of Acute Lower Limb Ischaemia : (Re-Open Registry)
Brief Title: Acute Limb Ischaemia (ALI) Management With 'Indigo' Mechanical Aspiration System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lancashire Care NHS Foundation Trust (Network)
Collaborators: St. Franziskus Hospital (Other)
Responsible Party: Principal Investigator, Bella Huasen, Endovascular Interventional Consultant, Lancashire Care NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Indigo2017
Record Dates: First submitted 2017-09-06; First posted 2017-09-28 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Lower Limb Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Acute or Chronic clot (Other): If chronic clot, no intervention given via Indigo
  Interventions: Device: 'Indigo' Mechanical thrombectomy system

INTERVENTIONS:
Device: 'Indigo' Mechanical thrombectomy system — Removal of acute clot from the artery causing ischaemia, using the mechanical aspiration system by Penumbra Inc called "INDIGO"

SUMMARY:
International Multi-Centre registry recording comprehensive data on the use of 'Indigo' Mechanical thrombectomy system by Penumbra Inc for the removal of acute clot causing acute or critical limb ischaemia.

DETAILED DESCRIPTION:
A detailed registry has been designed and approved to be used world wide in vascular and trauma centres, already providing endovascular service for the management of critical limb ischaemia (CLI).

Recent campaigns have shown little is done to improve flow to the lower limbs (legs) of patients to avoid amputation rates. During this time many devises have been used and available on the market. The 'Indigo' system by Penumbra was originally designed from the acute stroke system "ACE". Similar principles were applied in designing the 'Indigo' system. This is currently being used in many centres to manage acute clot causing lower limb ischaemia, however no official registry or international clinical trial has been done to show its significance in managing this disease.

The investigator groups, have created this to come up with enough data to evaluate the Indigo system in the management of (ALI) and offer tips and tricks to other clinicians. The aim is for a single arm, multicenter, retrospective analysis of patients in whom (ALI) was performed with the Penumbra/Indigo System (study device), and gather greater data and information than the PRISM trial in 2013-2014 which obtained only 79 patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute lower limb Ischaemia with acute soft clot.

Exclusion Criteria:

* Calcified plaques/ chronic disease causing critical limb Ischaemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Technical success using the Indigo system. | Time to event anaylsis. Primary patency results are immediate after the case on the final angiogram images.
  Intraoperative technical success defined as the restoration of antegrade blood flow with complete or near complete (95% by volume) removal of the thrombus or embolus (70% threshold). This is assessed using imaging modalities (USS/Doppler/Fluroscopy) and clinical assessment of the affected limb.
  See for this definition the enclosed citation. In conclusion, the primary outcome measure will be improvement in blood flow across a lesion assessed by the improvement in Thrombolysis in Myocardial Infarction (TIMI) score that was adapted to peripheral arteries. Concomitant balloon angioplasty or stent placement in addition to VAT was considered a complementary treatment. Additional thrombectomy treatments, such as thrombolysis and mechanical thrombectomy, were considered technical failures.Target lesions were grouped anatomically into above-the-knee(ATK) or below-the-knee(BTK) lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Bella Huasen, MD, Study Chair — Lancashire NHS
Locations (1):
- Interventional Radiology, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The registry and data in-put
Supporting Information: Study Protocol
Time Frame: while the study is on-going
Access Criteria: Centres taking part will be given the access via the three main trial investigators Dr Huasen, Dr Bisdas, and Dr Beropoulis

REFERENCES:
- [Result] Karnabatidis D, Spiliopoulos S, Tsetis D, Siablis D. Quality improvement guidelines for percutaneous catheter-directed intra-arterial thrombolysis and mechanical thrombectomy for acute lower-limb ischemia. Cardiovasc Intervent Radiol. 2011 Dec;34(6):1123-36. doi: 10.1007/s00270-011-0258-z. Epub 2011 Sep 1. PMID 21882081